CLINICAL TRIAL: NCT07033195
Title: Efficacy of a Virtual Reality Neuroscience-based Therapy (VRNT) for Chronic Low Back Pain
Brief Title: Virtual Reality Treatment for Adults With Chronic Back Pain (VRNT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CognifiSense Inc. (Industry)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0138
Record Dates: First submitted 2025-06-06; First posted 2025-06-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Chronic Back Pain; Chronic Lower Back Pain (CLBP)
Keywords: chronic pain relief; back pain; chronic back pain; chronic lower back pain
MeSH Terms: conditions — Chronic Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Virtual Reality Neuropsychological Therapy (Experimental): Participants start the treatment period with three introductory sessions:
  1. A 34-minute pain education video that introduces the neuroscience of acute and chronic pain, drivers of pain chronification, pain triggers, and the scientific principles behind the VRNT.
  2. A session to customize the VR experience to match the participant's experience using a display of a personalized 3-dimensional audiovisual representation of each patient's pain.
  3. A training session on the use of the VR hardware. The participant will receive a workbook to guide them through each day's session.
  Participants may continue their other pain treatment regimes, and are asked to notify the research team of any changes.
  Interventions: Device: Skills-based Virtual Reality Therapy
- Virtual Reality Neuroscience Therapy (Active Comparator): Participants start the treatment period with two introductory sessions: 1. A 7-minute pain education video that introduces the neuroscience of pain-focused attention, distraction, and the scientific principles behind VRNT. 2. A training session on the use of the VR hardware. The participant will receive a workbook (Attachment 'VRNT Workbook') to guide them through each day's session. Participants may continue their other pain treatment regimes, and are asked to notify the research team of any changes.
  Interventions: Device: Distraction-based Virtual Reality Therapy

INTERVENTIONS:
Device: Skills-based Virtual Reality Therapy — 1. A 34-minute education video session on the science behind chronic pain and the scientific principles of the therapy.
  2. VR skills-based therapy: a virtual reality therapy consisting of different psychological training exercises
  Arms: Virtual Reality Neuropsychological Therapy
Device: Distraction-based Virtual Reality Therapy — 1. A 7-minute education video session on the science behind pain-focused attention and distraction. 2. VR distraction-based therapy: a virtual reality therapy that encourages passive attention and minimizes external cognitive demands.
  Arms: Virtual Reality Neuroscience Therapy

SUMMARY:
Participants with chronic back pain will complete an online Qualtrics eligibility survey. After signing a consent form, eligible participants enter a two-week baseline period ("Baseline Period"), during which they complete two assessments of the Primary and Secondary Outcome Measures and Potential Mediators. After the baseline period, participants are randomized into a Virtual Reality group: VR Distraction-based Therapy or VR Skills-based Therapy, with a 1:1 allocation ratio of participants to each treatment. Both groups receive education on pain neuroscience and complete training on the use of the VR hardware and software. Next, both groups complete an intervention for 8 weeks ("Treatment Period"), after which they return the VR equipment. Several surveys are administered online during the Treatment Period. After the Treatment Period, both groups complete three post-treatment surveys at weeks 8, 20, and 32.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 85.
* Self-reported diagnosis of chronic low back pain without radicular symptoms.
* Chronic low back pain duration of 6 months or more, and pain at least half the days in the last 6 months.
* Lower back pain as primary chronic pain complaint (greater than pain in other bodily regions).
* Average pain intensity of 4 or more out of 10 for the past week (from BPI-SF).
* English fluency (8th grade level).
* Willing to comply with study procedures/restrictions.
* Access to Wi-Fi.
* Implicit de facto internet and computer literacy.

Exclusion Criteria:

* Applicants, who are pregnant, planning pregnancy, or breastfeeding
* Back pain associated with compensation / litigation within 1 year.
* Leg pain greater than back pain (suggests neuropathic pain; may be less responsive to psychological therapy).
* Chronic pain other than chronic back pain.
* Diagnoses of schizophrenia, multiple personality dissociative identity disorder.
* History of major depressive disorder not controlled with medication or other conditions that produce significant cognitive or emotional disability.
* History of substance abuse.
* Inability to undergo MRI (determined at screening; see XVI: Risks to Participants).
* Any clinically significant unstable medical abnormality or acute or chronic disease of cardiovascular, gastrointestinal, respiratory (e.g., chronic obstructive pulmonary disease), hepatic, or renal systems; including: history of cardiovascular disease or issues (e.g., recent heart attack), stroke; brain surgery, or brain tumor; Diabetes; cancer (last 12 months); diagnosis of a specific inflammatory disorder: rheumatoid arthritis, polymyalgia rheumatica, scleroderma, Lupus; polymyositis; or Cauda Equina syndrome.
* History of seizure disorder, epilepsy, convulsions, or increased intracranial pressure anytime except pediatric febrile seizures.
* History of vertigo, dizziness, susceptibility to motion sickness
* History of head injury within 6 months,
* Unexplained, unintended weight loss of 'â• 20 lbs in past year. Self-reported history of (digital) eye strain or computer vision syndrome. Unable or unwilling to meet study attendance requirements. MRI contraindications as determined by MRI safety screen (e.g., pregnancy, metal in body, claustrophobia, using the standard screen conducted by the MRI imaging facility).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity and Interference | Change from pre-treatment to post-treatment = 8 weeks
  Brief Pain Inventory-short form (BPI-SF). Measured on a Scale of 0 to 10, 0 = no pain, 10 = worst pain imaginable.

SECONDARY OUTCOMES:
Pain Interference | Change from pre-treatment to post-treatment = 8 weeks
  Brief Pain Inventory-short form (BPI-SF). Measured on a Scale of 0 to 10, 0 = no interference, 10 = severe interference.
Disability | Change from pre-treatment to post-treatment = 8 weeks
  Oswestry Low Back Pain Disability Questionnaire (OLBPQ). Measured on a scale of 0-100%, 0-20% = minimal disability, 80-100% = patients are bed-bound or exaggerating symptoms.
Physical Function | Change from pre-treatment to post-treatment = 8 weeks
  Physical Function (PROMIS). 5-point Likert scale: 5 = without any difficulty, 1 = unable to do (worse outcome).
Sleep Disturbance | Change from pre-treatment to post-treatment = 8 weeks
  Sleep Disturbance (PROMIS). 5-point Likert scale: 1 = very good, 5 = very poor (worst outcome).
Depression | Change from pre-treatment to post-treatment = 8 weeks
  Depression (PROMIS). 5-point Likert scale: 1 = never, 5 = always (worst outcome).
Anxiety | Change from pre-treatment to post-treatment = 8 weeks
  Anxiety (PROMIS). 5-point Likert scale: 1 = never, 5 = always (worst outcome).
Fatigue | Change from pre-treatment to post-treatment = 8 weeks
  Fatigue (PROMIS). 5-point Likert scale: 1 = not at all, 5 = very much (worst outcome).
Stress | Change from pre-treatment to post-treatment = 8 weeks
  Perceived Stress Scale (PSS). Measured on a scale of 0 to 40, 0-13 = low stress, 27-40 = high perceived stress.

OTHER OUTCOMES:
Cybersickness | Assessed at Week 8
  Single item questionnaire: "Did you experience any motion sickness or nausea while using VR?". 4-point Likert Scale: 0 = never, 3 = always (worst outcome).
Global Improvement | Assessed at Week 8
  Patient's Global Impression of Change (PGIC). 10-point Likert scale: 0 = much better, 10 = much worse (worst outcome).
Treatment Satisfaction | Assessed at Week 8
  Treatment satisfaction (single item). 7-point Likert scale: extremely satisfied, extremely dissatisfied (worst outcome).
System Usability | Assessed at Week 8
  System usability (SUS). 5-point Likert scale: 1 = strongly disagree, 5 = strongly agree.
Virtual Reality Device Use | Throughout treatment = 8 weeks
  Data collected from VR Device
Chronic Pain Acceptance | Change from pre-treatment to post-treatment = 8 weeks
  Chronic Pain Acceptance Questionnaire (CPAQ-8). 7-point Likert scale: 6 = always true, 0 = never true (worst outcome).
Pain catastrophizing | Change from pre-treatment to post-treatment = 8 weeks
  Pain catastrophizing (PCS). 5-point Likert scale: 0 = not at all, 4 = all the time (worst outcome).
Pain self-efficacy | Change from pre-treatment to post-treatment = 8 weeks
  Pain Self-Efficacy Questionnaire (PSEQ-2). 7-point Likert scale: 6 - completely Confident, 0 = not at all confident (worst outcome).
Positive and Negative affect | Change from pre-treatment to post-treatment = 8 weeks
  Positive and Negative Affect Schedule (PANAS-SF). 5-point Likert scale: 1 = very slightly, 5 = extremely.
Fear of movement | Change from pre-treatment to post-treatment = 8 weeks
  Tampa Scale Kinesiophobia (TSK). 4-point Likert scale: 1 = strongly disagree, 4 - strongly agree (worst outcome).
Immersive tendencies | Change from pre-treatment to post-treatment = 8 weeks
  Immersive Tendencies Questionnaire (ITQ). 7-point Likert scale: never, often.
Expectations of treatment success | Change from pre-treatment to post-treatment = 8 weeks
  Expectations of Treatment Success. 10-point Likert scale: 10 = most, 0 = none.
Adherence | Throughout treatment = 8 weeks
  Data collected from VR Device
Medication Use | Change from pre-treatment to post-treatment = 8 weeks
  Custom analgesic medication use survey. Data collection of medication type, frequency of use, and dose standardized with "Opioid Oral Morphine Milligram Equivalent (MME) Conversion Table"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Landing Page for the study — https://studies.buildclinical.com/bcfs001533-cu-ceko-84-landing-page/